CLINICAL TRIAL: NCT04970797
Title: Using EEG and Metabolomics to Evaluate the Clinical Efficacy of Xinglouchengqi Decoction in Improving Nerve Injury in the Acute Stage of Stroke and the Mechanism
Brief Title: Mechanism of Xinglouchengqi Decoction in Improving Nerve Injury in the Acute Stage of Stroke by EEG and Metabolomics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Xin Xiyan, Attending physician, Peking University Third Hospital
Other Study IDs: M2019430
Record Dates: First submitted 2021-07-02; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional treatment group: Western medicine treatment
- Combination treatment group: Xinglouchengqi decoction combined with western medicine treatment
  Interventions: Drug: Xinglouchengqi decoction

INTERVENTIONS:
Drug: Xinglouchengqi decoction — the composition of Xinglouchengqi decoction: 9 g raw rhubarb, 9 g mirabilite, 6 g dananxing, 30 g quangualou decoction was uniformly prepared by the pharmacy department of our hospital. Decoction form was adopted, one dose per day, one dose of 200 mL decoction, and the decoction was taken in morning and evening twice and half an hour after meals. The observation period was 5 days: from 72 hours to 7 days after onset.
  Other Names: 9 g raw rhubarb, 9 g mirabilite, 6 g dananxing, 30 g quangualou decoction
  Groups: Combination treatment group

SUMMARY:
Using EEG and metabolomics to evaluate the clinical efficacy of Xinglouchengqi decoction in improving nerve injury in the acute stage of stroke and the mechanism

DETAILED DESCRIPTION:
Traditional Chinese medicine treatment is the original advantage in China for early stroke intervention. Xinglouchengqi decoction is an important prescription for the treatment of acute stage of stroke proposed by Academician Wang Yongyan. Early intervention can significantly improve the condition of patients and reduce the degree of neurological function deficit, but its mechanism of action is not clear.EEG, network graph theory and metabonomics are applied in evaluating the treatment of stroke, and to explore the mechanism of Xinglouchengqi decoction to improve the nerve injury of acute stroke patients. 30 stroke patients with acute period will be as the research object, using the observational cohort studies, to measure the dynamic of nerve function defect, EEG signals and other clinical information. Based on EEG to construct the brain functional network in the acute stage of stroke and to study the brain network mechanism of Xinglouchengqi decoction in improving the nerve injury of patients. Meanwhile, based on the study of metabolomics, the potential biomarkers and the metabolic pathway will be analyse to explore the pharmacodynamic substance.

ELIGIBILITY:
Inclusion Criteria:

those who met the diagnostic criteria for acute anterior circulation ischemic stroke; first stroke, no previous history of organic encephalopathy; the onset is less than 72 hours; it is in line with the TCM diagnosis of phlegm heat; aged 40 to 80 years old.

Exclusion Criteria:

Transient Ischemic Attack (TIA) ; those who have received thrombolytic therapy; the examination confirmed that the stroke was caused by the brain tumor, brain trauma or blood disease; cerebral embolism caused by rheumatic heart disease, coronary heart disease and other heart disease combined with atrial fibrillation; complicated with liver and kidney hematopoietic system endocrine system and other serious diseases and osteoarthropathy; prior mental disorder or severe dementia; patients with concurrent infection and fever; patients with primary or secondary epilepsy; those who had taken sedative drugs or sleeping drugs 3 days before the examination.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: those who met the diagnostic criteria for acute anterior circulation ischemic stroke; first stroke, no previous history of organic encephalopathy; the onset is less than 72 hours; it is in line with the TCM diagnosis of phlegm heat; aged 40 to 80 years old.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
parameters of EEG | Within 72 hours of onset
  Brain network parameters based on EEG
parameters of EEG | Day 5
  Brain network parameters based on EEG
parameters of EEG | Day 7
  Brain network parameters based on EEG
LC-MS results | Within 72 hours of onset
  To explore the possible biomarkers, metabolic pathways, metabolic networks using blood and urine samples
LC-MS results | Day 5
  To explore the possible biomarkers, metabolic pathways, metabolic networks using blood and urine samples
LC-MS results | Day 7
  To explore the possible biomarkers, metabolic pathways, metabolic networks using blood and urine samples
NIHSS | Within 72 hours of onset
  Stroke Scale NIHSS
NIHSS | day 5
  Stroke Scale NIHSS
NIHSS | day 7
  Stroke Scale NIHSS
BI scale | day 30
  To assess the activity of daily living scale Barthel Index (BI)
mRS scale | day 30
  Modified Rankin Scale (mRS)
Head MRI | Within 72 hours of onset
  The location and size of the lesions were recorded in detail

IPD SHARING:
Plan to Share IPD: No